CLINICAL TRIAL: NCT05375058
Title: Impact of the COVID-19 Pandemic on the Incidence of Complicated Appendicitis in a Tertiary Medical Center, Amman, Jordan: A Retrospective Cohort
Brief Title: Complicated Appendicitis During the COVID-19 Pandemic in Jordan
Status: Completed | Type: Observational
Sponsor: Jordan University Hospital (Other)
Responsible Party: Principal Investigator, Abdallah Raed Al-Qawasmeh, Co-Principal Investigator, Jordan University Hospital
Other Study IDs: 28/2021
Record Dates: First submitted 2022-05-11; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: COVID-19; Complicated Appendicitis
MeSH Terms: conditions — COVID-19 | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pandemic group (2020): includes patients who presented to the hospital during the period of acute restrictions and shutdowns extending from the 17th of March to the 6th of June 2020
  Interventions: Other: Observational Study
- pre-pandemic group (2019): which represents the same period in the previous year

INTERVENTIONS:
Other: Observational Study — Observational Study; the study did not involve any interventions
  Groups: pandemic group (2020)

SUMMARY:
Comparing the incidence of complicated appendicitis between two groups, the pandemic and pre-pandemic groups.

DETAILED DESCRIPTION:
The investigators have retrospectively investigated data on acute appendicitis cases. Two groups were established, the first group was the pandemic group, which included patients who presented to the hospital during the period of acute restrictions and shutdowns extending from the 17th of March to the 6th of June 2020, and the pre-pandemic group which represents the same period in the previous year, the aim was to assess the incidence of complicated appendicitis during the COVID-19 pandemic in Jordan University Hospital

ELIGIBILITY:
Inclusion Criteria:

* Any patient that presented with appendicitis and underwent an appendectomy at the university of Jordan hospital during the specified time periods (March 2019-December 2020)

Exclusion Criteria:

* Incomplete data record.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient that has a medical record for appendicitis and underwent appendectomy at University of Jordan hospital
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2019-03-02 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Occurrence of postoperative complications | Up to 2 years
  To determine if there were any complications, this was detected by reviewing the histopathology report

SECONDARY OUTCOMES:
Length of in-hospital stay | Up to 2 years
  How many days did the patient spend in the hospital until discharged.
Imaging method used for diagnosis (CT or US) | Up to 2 years
  How was appendicitis diagnosed, either by using Computed Tomography (CT) Scan or Ultrasound.
Type of operation (open or laparoscopic) | Up to 2 years
  We reported what type of operation the patient underwent to treat appendicitis.

CONTACTS AND LOCATIONS:
Overall Officials: Marzouq Amarin, MD, MSc, Principal Investigator — Department of General Surgery, the University of Jordan, Amman, 11942, Jordan
Locations (1):
- Jordan University Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided